CLINICAL TRIAL: NCT06231563
Title: Examining Ketamine Effects on Depression, Neuroplasticity, and Inflammation in Veterans With Parkinson's Disease
Brief Title: Ketamine for Veterans With Parkinson's Disease
Acronym: KPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBC-004-23S; 23-40158 (Other: UCSF Institutional Review Board (IRB)); CX002606 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Ketamine; Depression; Inflammatory markers; Neuroplasticity; Clinical Trial Protocol
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Ketamine; remimazolam

STUDY DESIGN:
Intervention Model Description: Veterans with Parkinson's disease (N=80) will be randomized to complete a single IV ketamine infusion or active placebo infusion (remimazolam).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-masked, active placebo-controlled, single dose randomized trial of intravenous (IV) ketamine for depression in people with Parkinson's disease (PD).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine (Experimental): intravenous ketamine infusion 0.5 mg/kg
  Interventions: Drug: Ketamine
- Remimazolam (Placebo Comparator): intravenous remimazolam infusion 0.25 mg/kg
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Ketamine — intravenous ketamine infusion 0.5 mg/kg
  Arms: Ketamine
Drug: Remimazolam — intravenous remimazolam infusion 0.25 mg/kg
  Arms: Remimazolam

SUMMARY:
Parkinson's disease (PD) is a devastating illness that has a growing impact on Veterans. One of the most disabling symptoms is depression, which is common in PD and linked to poor quality of life and higher risk of suicide. Unfortunately, there is a lack of effective treatments for depression in PD. Ketamine, which has rapid and potent antidepressant effects, is a potential option but has not been tested in Veterans with PD. Studies in rodents show that ketamine may not only improve depression in PD, it may target two of the underlying drivers of the disease: (1) reduced neuroplasticity, or the brain's ability to adapt and remodel itself; and (2) elevated inflammation. The investigators are conducting a randomized, placebo-controlled study to examine if a dose of intravenous (IV) ketamine improves depression in Veterans with PD. The investigators will also examine ketamine's effects on neuroplasticity and inflammation, which will help us understand how ketamine works in PD and if it can be a useful treatment for Veterans with the disease. This study will lay groundwork for a larger clinical trial across multiple VA sites.

DETAILED DESCRIPTION:
This is a double-masked, active placebo-controlled, single dose randomized trial of intravenous (IV) ketamine versus remimazolam for depression in Veterans (N=80) with Parkinson's disease (PD). The investigators hypothesize that ketamine will have a strong safety and tolerability profile and improve depressive symptoms within 24 hours (Aim 1). Further, its antidepressant effects will be associated with modulation of both impaired neuroplasticity (Aim 2) and elevated inflammatory activity (Aim 3). To test these hypotheses, the investigators will use clinical assessments (of adverse events, tolerability, and depression), non-invasive brain stimulation techniques to quantify changes in LTP-like neuroplasticity, and blood-based cytokine measurement to quantify changes in systemic inflammation. This study will provide clinical efficacy data and elucidate ketamine's mechanisms of action in PD using accessible, neuroscience-informed markers of neuroplasticity and inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide written informed consent.
2. Is a United States Veteran.
3. Between 40-80 years old at the time of informed consent
4. Have neurologist-diagnosed idiopathic Parkinson's disease (PD) for at least six months prior to enrollment
5. History of inadequate response to at least one trial of antidepressant medication
6. On a stable regimen of all medications for at least 2 months prior to enrollment and have no planned medication changes during the period of active participation.
7. Commit to attend all in-person and remote study visits and participate in all data collection procedures.
8. Have a score >/=20 on the Montgomery-Asberg Depression Rating Scale (MADRS), consistent with moderate or greater depressive symptom severity, at Baseline.
9. If already engaged in psychotherapy or other non-pharmacologic treatments for depression, agree to maintain consistent engagement throughout the period of active study participation.
10. If not engaged in psychotherapy or other non-pharmacologic treatments for depression, agree to avoid starting a new course of treatment for the period of active study participation.
11. Agree to abstain from cannabis for a minimum of 72 hours prior to assessments on Day - 1 and to remain abstinent through assessments on Day 0
12. If a regular user of tobacco or nicotine, agree to maintain a consistent pattern of use throughout the period of active study participation; if an infrequent/occasional user, agree to abstain throughout the period of active study participation
13. For people who can become pregnant or trying to conceive: agree to use highly effective contraception from entry into the trial through Day 7 assessments

Exclusion Criteria:

1. Lifetime history of schizophrenia or schizoaffective disorder or bipolar disorder or current psychosis with loss of insight
2. Dementia or cognitive impairment as determined by a MoCA (telephone version) score <18 at screening.
3. Moderate or severe substance use disorder during the 6 months prior to enrollment or a breathalyzer test showing an alcohol level > 0% at screening or a positive urine toxicology panel at screening. Note that a positive result for cannabis is an exception; see Inclusion Criteria
4. Pregnancy, breastfeeding, or plans to become pregnant during the period of trial participation.
5. Electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) treatment within 30 days prior to enrollment or plans to begin either therapy during the participation period
6. High risk of self-harm/suicide that warrants immediate treatment as determined by the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening
7. Current severity of depression symptoms warranting immediate treatment (i.e., resulting in inability to provide for basic needs/safety) at screening
8. Meeting standard safety exclusion criteria for TMS (seizure disorder, ferrous metal or implanted devices above the chest, history of severe traumatic brain injury, tinnitus)
9. Meeting standard safety exclusion criteria for ketamine treatment (previous hypersensitivity reaction to ketamine, hepatitis or liver failure, cystitis, or underlying cardiovascular conditions in which increased blood pressure would pose a risk of complications)
10. Concomitant medications that may interfere with ketamine treatment or increase risk of adverse events (e.g., benzodiazepines, sedative-hypnotics, lamotrigine, MAOIs) if it is not medically appropriate or feasible for the participant to abstain from use for at least 5 half-lives prior to assessments on Day -1 and remain abstinent through assessments on Day 0
11. Concomitant medications that may impact motor cortex plasticity (e.g., memantine, dextromethorphan) if it is not medically appropriate or feasible for the participant to abstain from use for at least 5 half-lives prior to assessments on Day -1 and remain abstinent through assessments on Day 0
12. Concomitant medications that may increase risk of adverse events with TMS (i.e,. those that can lower the seizure threshold) if it is not medically appropriate or feasible for the participant to abstain from use for at least 5 half-lives prior to assessments on Day -1 and remain abstinent through assessments on Day 0
13. Autoimmune disorders (e.g., multiple sclerosis, lupus, rheumatoid arthritis) or neoplastic disorders
14. Use of cytokine antagonists or other medications that may modulate inflammation unless regimen has been stable for at least 2 months and there is no plan to alter the regimen during trial participation
15. Another medical condition or diagnosis, physical exam finding, or laboratory abnormality that precludes participation in study procedures due to safety concerns.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | baseline and 24 hours post-infusion.
  Changes in depression as measured by the Montgomery-Asberg Depression Rating Scale (MADRS) between baseline and 24 hours post-infusion. Overall score ranges from 0 to 60, where higher scores indicate more severe depression

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline to 24 hours post-infusion, Day 3, Day 5, Day 7
  Changes in depression severity as measured by Montgomery-Asberg Depression Rating Scale scores. Overall score ranges from 0 to 60, where higher scores indicate more severe depression
Hamilton Depression Rating Scale-7 (HAMD-7) | Baseline to 24 hours post-infusion, Day 3, Day 5, Day 7
  Changes in core depressive symptoms as measured by the Hamilton Depression Rating Scale-7. Overall score ranges from 0 to 56, where higher scores indicate more severe depression
Patient- Reported Outcomes Measurement Information System (PROMIS®) | Baseline to Day 7
  Changes in functional impairment related to PD as measured by the Patient- Reported Outcomes Measurement Information System (PROMIS®), where higher scores indicate more impairment
Quality of Life in Neurological Disorders (Neuro-QoLTM) | Baseline to Day 7
  Changes in quality of life measured by select measures on the Quality of Life in Neurological Disorders (Neuro-QoLTM), where higher scores indicate more impairment
Incidence, severity, and frequency of Adverse Events (AEs) including Treatment- Emergent AEs (TEAEs) and Serious AEs (SAEs) | Baseline to Day 7
  Incidence, severity, and frequency of Adverse Events (AEs) including Treatment- Emergent AEs (TEAEs) and Serious AEs (SAEs)
Ketamine Side Effect Tool (KSET) | Baseline to Day 7
  Incidence, severity and frequency of AEs using a study-specific adaptation of the Ketamine Side Effect Tool (KSET)
Enhanced Scale for the Assessment of Positive Symptoms for Parkinson's Disease (eSAPS- PD) | Baseline to Day 7
  Changes in clinician-rated psychotic symptoms assessed using the Enhanced Scale for the Assessment of Positive Symptoms for Parkinson's Disease (eSAPS- PD). Scores range from 25 to 125, where higher scores indicate more impairment
Frequency, Intensity, Burden of Side Effects Rating Scale (FIBSER) | Day 7
  Tolerability as assessed by the Frequency, Intensity, Burden of Side Effects Rating Scale (FIBSER). Scores range from 0-6, where higher scores indicate more impairment
Hamilton Anxiety Rating Scale (HAM-A) | Baseline to 24 hours post-infusion, Day3, Day 7
  Changes in anxiety as measured by the Hamilton Anxiety Rating Scale (HAM-A); Overall score ranges from 0 to 56, where higher scores indicate more severe anxiety
Movement Disorder Society revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline to 4 hours post-infusion, 24 hours post-infusion, Day 3, Day 5, Day 7
  Changes in PD symptom severity measured by the Movement Disorder Society revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
transcranial magnetic stimulation (TMS) | Baseline to 4 hours post-infusion
  Changes in brain structure as measured by transcranial magnetic stimulation (TMS)
Changes in inflammatory index as measured by blood-based analysis | Baseline to 4 hours post-infusion
  Changes in inflammatory index as measured by blood-based analysis
transcranial magnetic stimulation (TMS) | Baseline to 4 hours post-infusion
  Changes in brain function as measured by transcranial magnetic stimulation (TMS)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Bradley, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No